CLINICAL TRIAL: NCT00375973
Title: A Randomized, Placebo-Controlled, Double-Blind Trial of Duloxetine in the Treatment of Patients With Chronic Fatigue Syndrome
Brief Title: Double Blind Trial of Duloxetine in Chronic Fatigue Syndrome
Acronym: CFS
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: University of Cincinnati (Other)
Collaborators: Eli Lilly and Company (Industry)
Responsible Party: Principal Investigator, Lesley M. Arnold, M.D., Professor, University of Cincinnati
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 06-05-01-02
Record Dates: First submitted 2006-09-12; First posted 2006-09-13 (Estimated); Results first posted 2015-07-27 (Estimated); Last update posted 2015-08-21 (Estimated); Status verified 2015-07

CONDITIONS: Fatigue Syndrome, Chronic
Keywords: Fatigue; Fatigue syndrome, chronic; Chronic fatigue syndrome; CFS; Fibromyalgia
MeSH Terms: conditions — Fatigue Syndrome, Chronic; Fatigue; Fibromyalgia | interventions — Duloxetine Hydrochloride; Sugars

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Duloxetine (Experimental): Duloxetine po 60-120 mg/day for 12 weeks
  Interventions: Drug: Duloxetine
- Placebo (Placebo Comparator): Placebo comparator to Duloxetine
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Duloxetine — Duloxetine po 60-120 mg/day for 12 weeks
  Other Names: Cymbalta
  Arms: Duloxetine
Drug: Placebo — Sugar pill dose comparable to duloxetine
  Other Names: Sugar Pill
  Arms: Placebo

SUMMARY:
The purpose of this study is to determine the safety and efficacy of duloxetine compared with placebo for reducing fatigue in patients diagnosed with Chronic Fatigue Syndrome (CFS).

DETAILED DESCRIPTION:
Chronic fatigue syndrome (CFS) is characterized by severe disabling fatigue of at least six months duration that cannot be fully explained by an identifiable medical condition . Pain symptoms are also a part of the diagnostic criteria for CFS, and include muscle pain, multi-joint pain, and headaches. The prevalence of CFS ranges from 0.007 to 2.8 % in the general adult population and 0.006 to 3.0% in primary care practice (2). Although most who receive a CFS diagnosis are 30-40 years of age, Caucasian, and female, CFS affects both women and men, adults and children, and all racial and socioeconomic classes.

Patients with CFS have 2-4 times the rate of depression and anxiety compared with the general population. CFS is also commonly comorbid with fibromyalgia, a disorder characterized by chronic widespread pain, tenderness, fatigue, sleep and mood disturbances. In some samples, 70% of patients with fibromyalgia also meet criteria for CFS. CFS and fibromyalgia are characterized by greater similarities than differences and may share pathophysiologic features. Like fibromyalgia, CFS is associated with chronic pain, sleep and mood disturbances. Because fibromyalgia responds to treatment with antidepressants, particularly the dual serotonin and norepinephrine reuptake inhibitors, including duloxetine, antidepressant trials in CFS are clearly needed.

ELIGIBILITY:
Inclusion Criteria:

1. Female and male outpatients between 18-65 years of age.
2. Meet criteria for revised Center for Disease Control (CDC) definition of Chronic Fatigue Syndrome (CFS) (at least 6 months of persistent fatigue that substantially reduces the person's level of activity; 4 or more of the following symptoms that must occur with fatigue in a 6-month period: impaired memory or concentration, sore throat, tender glands, aching or stiff muscles, multijoint pain, new headaches, unrefreshing sleep, and post-exertional fatigue. Medical conditions that may explain the fatigue and psychiatric disorders, including eating disorders, psychotic disorders, bipolar disorder, melancholic depression, and substance abuse within 2 years of the onset of fatigue, are excluded).
3. Provision of written informed consent for participation in the trial.
4. Educational level and degree of understanding such that the patient can communicate intelligibly with the investigator and study staff.
5. Judged to be reliable and agree to keep all appointments for clinic visits, tests, and procedures required by the protocol.

Exclusion Criteria:

1. Current melancholic major depressive disorder, or a previous diagnosis of psychosis, eating disorder, or bipolar disorder.
2. History of substance abuse or dependence within the past year, excluding nicotine and caffeine.
3. A positive urine drug screen for any substance of abuse (may be retested if positive test was for a prescribed medication that was not washed out).
4. Women who are pregnant or breast feeding; women must test negative for pregnancy at Visit 1.
5. Women of childbearing potential who are not using a medically accepted means of contraceptive when engaging in sexual intercourse.
6. Patients who, in the opinion of the investigator, are treatment-refractory or whose response is likely to be compromised by existing or future disability compensation issues.
7. Serious unstable medical illness, including cardiovascular, hepatic, renal, respiratory, or hematologic illness, or other unstable medical or psychiatric conditions that in the opinion of the investigator would compromise participation or would likely lead to hospitalization during the duration of the study. Abnormal thyroid stimulating hormone (TSH) concentrations (unless treatment for hypothyroidism has been stable for at least the past 3 months and the patient is clinically euthyroid).
8. Patients who have uncontrolled narrow-angle glaucoma.
9. Patients who have acute liver injury (such as hepatitis) or severe cirrhosis (Child-Pugh Class C).
10. Patients who are judged prior to randomization to be at suicidal risk by the clinical investigator.
11. Treatment with antidepressant medication within 14 days prior to randomization with the exception of fluoxetine, which cannot be used within 30 days prior to randomization. Potential need to use a monoamine oxidase inhibitor (MAOI) during the study or within 2 weeks of discontinuation of study treatment.
12. Patients who have previously taken duloxetine
13. Patients who are taking any excluded medications that cannot be discontinued at Visit 1.
14. Treatment within the last 30 days with a drug that has not received regulatory approval at the time of study entry.
15. Known hypersensitivity to duloxetine or any of the inactive ingredients.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2006-09; Primary Completion 2012-06 (Actual); Study Completion 2014-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lesley M Arnold, MD, Principal Investigator — University of Cincinnati Women's Health Research Program
Locations (1):
- Women's Health Research Program, Cincinnati, Ohio, United States

REFERENCES:
- [Derived] Arnold LM, Blom TJ, Welge JA, Mariutto E, Heller A. A randomized, placebo-controlled, double-blinded trial of duloxetine in the treatment of general fatigue in patients with chronic fatigue syndrome. Psychosomatics. 2015 May-Jun;56(3):242-53. doi: 10.1016/j.psym.2014.12.003. Epub 2014 Dec 16. PMID 25660434

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Duloxetine | Placebo
Started | 30 | 30
Completed | 20 | 28
Not Completed | 10 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Duloxetine | Placebo | Total
Number analyzed (Participants) | 30 | 30 | 60
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 30 | 30 | 60
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 43.0 (11.8) | 44.3 (11.0) | 43.6 (11.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 26 | 26 | 52
  Male | 4 | 4 | 8
Region of Enrollment [Number; unit: participants]
  United States | 30 | 30 | 60

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Multidimensional Fatigue Inventory (MFI)--General Fatigue Subscale Score
Description: The MFI is a self-reported instrument that contains 20 statements covering different aspects of fatigue. The MFI consists of 5 subscales: general fatigue, physical fatigue, mental fatigue, reduced activity, and reduced concentration. Each subscale includes 4 items with 5-point Likert scales. Scores on each subscale range from 4-20 with higher scores indicating greater fatigue. A decrease in the score indicates improvement.
  The general fatigue subscale (primary measure) includes general statements about tiredness, feeling rested, and overall feelings of being fit.
Time Frame: Baseline to endpoint at 12 weeks
Population: For the efficacy analysis, in the duloxetine group, 3 patients were not included in analysis for the following reasons: one patient's treatment group assignment was unblinded owing to a serious adverse event of suicidal ideation; 2 other patients did not have compliant postbaseline visits.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Duloxetine | Placebo
Number analyzed (Participants) | 27 | 30
units on a scale | -3.3 (4.2) | -1.8 (2.8)
Statistical Analysis 1: Comparison: Duloxetine vs Placebo; Test type: Superiority or Other; p = 0.23, Regression, Linear

2. Secondary Outcome: Change From Baseline in Brief Pain Inventory (BPI) --Average Pain Severity Score
Description: The BPI is a self-administered scale that measures the severity of pain. Pain severity is rated on a 0 [no pain] to 10 [pain as bad a you can imagine] scale. Average pain is rated over the previous 24 hours. Higher scores indicate greater pain severity. A decrease in the score indicates improvement (i.e. decrease in pain severity).
Time Frame: Baseline to endpoint at 12 weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Duloxetine | Placebo
Number analyzed (Participants) | 27 | 30
units on a scale | -1.6 (1.5) | -0.8 (2.3)
Statistical Analysis 1: Comparison: Duloxetine vs Placebo; Test type: Superiority or Other; p = 0.05, Regression, Linear

3. Secondary Outcome: Change From Baseline in the Hospital Anxiety and Depression Scale (HADS) --Depression Subscale
Description: The HADS is a self-reported instrument designed as a brief assessment tool of anxiety and depression in nonpsychiatric populations. It is a 14-item questionnaire that consistes of 2 subscales of 7 items designed to measure levels of both anxiety and depression. Each item on the questionnaire is scored from 0-3 and this means that a person can score between 0 and 21 for either anxiety or depression. Higher scores indicate greater levels of anxiety or depression. A decrease in the score indicates improvement.
Time Frame: baseline to endpoint at 12 weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Duloxetine | Placebo
Number analyzed (Participants) | 27 | 30
units on a scale | -1.6 (2.9) | -1.9 (3.0)
Statistical Analysis 1: Comparison: Duloxetine vs Placebo; Test type: Superiority or Other; p = 0.67, Regression, Linear

4. Secondary Outcome: Change From Baseline in the Clinical Global Impression of Severity (CGI-S)
Description: Clinician rated assessment of severity on a 1 (normal)-7 (extremely ill) scale. A decrease in the score indicates improvement.
Time Frame: baseline to endpoint at 12 weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Duloxetine | Placebo
Number analyzed (Participants) | 27 | 30
units on a scale | -1.1 (1.2) | -0.4 (1.0)
Statistical Analysis 1: Comparison: Duloxetine vs Placebo; Test type: Superiority or Other; p = 0.02, Regression, Linear

5. Secondary Outcome: Patient Global Impression of Improvement (PGI-I)
Description: Patient rated assessment of change on a 1 (very much better) to 7 (very much worse) scale.
Time Frame: baseline to endpoint at 12 weeks.
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Duloxetine | Placebo
Number analyzed (Participants) | 27 | 30
units on a scale | 3.2 (1.2) | 3.3 (1.2)
Statistical Analysis 1: Comparison: Duloxetine vs Placebo; Test type: Superiority or Other; p = 0.06, Regression, Linear

6. Secondary Outcome: Number of Participants Who Discontinued the Study for Any Reason
Description: Description of discontinuation rates of participants; all participants who dropped out of the study after randomization were included. The reasons for drop outs included lack of efficacy, adverse event, lost to follow-up, personal conflict or other patient decision, withdrawal of informed consent, and non-compliance.
Time Frame: Any time after randomization up to 12 weeks.
Measure: Number; unit: participants
Arm/Group | Duloxetine | Placebo
Number analyzed (Participants) | 30 | 30
participants | 10 | 2
Statistical Analysis 1: Comparison: Duloxetine vs Placebo; Test type: Superiority or Other; p = 0.02, Fisher Exact

7. Secondary Outcome: Number of Participants Who Discontinued Use of Treatment Due to Adverse Events
Description: Paticipants who dropped out of the study because of intolerable adverse events.
Time Frame: Any time after randomization up to 12 weeks.
Population: One patient in the duloxetine group did not have post-baseline data.
Measure: Number; unit: participants
Arm/Group | Duloxetine | Placebo
Number analyzed (Participants) | 29 | 30
participants | 3 | 0
Statistical Analysis 1: Comparison: Duloxetine vs Placebo; Test type: Superiority or Other; p = 0.24, Fisher Exact

ADVERSE EVENTS:
Arm/Group | Duloxetine | Placebo
Serious Adverse Events (participants affected / at risk) | 1/29 | 0/30
Other Adverse Events (participants affected / at risk) | 29/29 | 30/30
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Duloxetine (N=29) | Placebo (N=30)
Suicidal ideation (Psychiatric disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Duloxetine (N=29) | Placebo (N=30)
Nausea (Gastrointestinal disorders) | 19 | 6
Somnolence (Nervous system disorders) | 12 | 3
dizziness (Nervous system disorders) | 9 | 2
headache (Nervous system disorders) | 3 | 12
dry mouth (Gastrointestinal disorders) | 6 | 1
Insomnia (Psychiatric disorders) | 10 | 4
Constipation (Gastrointestinal disorders) | 8 | 5
Cold virus (Infections and infestations) | 5 | 7
Decreased appetite (Gastrointestinal disorders) | 5 | 1
Diarrhea (Gastrointestinal disorders) | 5 | 3
Lightheadedness (Nervous system disorders) | 5 | 3
Anxiety (Psychiatric disorders) | 4 | 1
Vivid dreams (Psychiatric disorders) | 4 | 1
Increased urination (Renal and urinary disorders) | 3 | 0
Increased yawning (Nervous system disorders) | 3 | 1
Jittery (Nervous system disorders) | 3 | 0
Increased sweating (Skin and subcutaneous tissue disorders) | 3 | 0
Chills (Skin and subcutaneous tissue disorders) | 2 | 0
Depression (Psychiatric disorders) | 2 | 1
Fever (Infections and infestations) | 2 | 0
Hot flush (Vascular disorders) | 2 | 0
Increased appetite (Gastrointestinal disorders) | 2 | 2
Irritabililty (Psychiatric disorders) | 2 | 4
Pruritus (Skin and subcutaneous tissue disorders) | 2 | 2
Muscle fasciculation (Musculoskeletal and connective tissue disorders) | 2 | 0
Abdominal pain (Gastrointestinal disorders) | 2 | 0
Sinus infection (Infections and infestations) | 2 | 2
Vaginal infection (Infections and infestations) | 2 | 1
Weight gain (Metabolism and nutrition disorders) | 2 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No